CLINICAL TRIAL: NCT00616031
Title: A Phase II, Multinational and Multicenter, Randomized, Controlled Study of Paclitaxel and Carboplatin With vs Without Nitroglycerin in Patients With Untreated Advanced Non-small Cell Lung Cancer
Brief Title: Paclitaxel and Carboplatin With or Without Nitroglycerin in Treating Patients With Previously Untreated Stage III or Stage IV Non-Small Cell Lung Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Kyoto University (Other)
Collaborators: Translational Research Center for Medical Innovation, Kobe, Hyogo, Japan (Other)
Organization: National Cancer Institute (NCI) (NIH)
Allocation: Randomized | Purpose: Treatment
Other Study IDs: TRIC-TRIL-C0702; CDR0000584254 (Registry Identifier: PDQ (Physician Data Query)); TRIC-C157
Record Dates: First submitted 2008-02-14; First posted 2008-02-15 (Estimated); Last update posted 2013-08-12 (Estimated); Status verified 2009-07

CONDITIONS: Lung Cancer
Keywords: stage IIIB non-small cell lung cancer; stage IV non-small cell lung cancer
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Non-Small-Cell Lung | interventions — Carboplatin; Nitroglycerin; Paclitaxel

INTERVENTIONS:
Drug: carboplatin
Drug: nitroglycerin
Drug: paclitaxel

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as paclitaxel and carboplatin, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Nitroglycerin may help carboplatin and paclitaxel work better by making tumor cells more sensitive to the drugs.

PURPOSE: This phase II randomized trial is studying how well giving nitroglycerin together with paclitaxel and carboplatin works and compares it to giving paclitaxel and carboplatin alone in treating patients with previously untreated stage III or stage IV non-small cell lung cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* To evaluate tumor response rate and safety of nitroglycerin as a potentiator of anticancer combination therapy comprising paclitaxel and carboplatin in patients with previously untreated stage IIIB or IV non-small cell lung cancer.

OUTLINE: This is a multicenter, randomized, controlled study. Patients are randomized to 1 of 2 treatment arms.

* Arm I: Patients receive nitroglycerin, paclitaxel, and carboplatin.
* Arm II: Patients receive paclitaxel and carboplatin. In both arms, treatment continues for 6 courses in the absence of disease progression or unacceptable toxicity.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically confirmed non-small cell lung cancer

  * Stage IIIB or IV disease that cannot be treated by radical irradiation
* Tumor lesions must be objectively evaluated according to WHO criteria (maximum diameter is no shorter than twice the slice width and no shorter than 10 mm) by CT scan
* No brain metastasis

PATIENT CHARACTERISTICS:

* ECOG performance status 0-1
* Life expectancy ≥ 3 months
* Neutrophil count > 2,000/μL
* Hemoglobin > 10.0 g/dL
* Platelet count > 100,000/μL
* Serum bilirubin < 2.0 mg/dL
* ALT and AST < 100 IU/L
* Serum creatinine < 2.0 mg/dL
* PaO_2 ≥ 70 mm Hg
* No cardiac problems, including any of the following:

  * Poorly controlled hypertension
  * Unstable angina
  * Congestive heart failure
  * Myocardial infarction within the past year
  * Ventricular arrhythmia that requires treatment except single, well-controlled isolated ventricular extrasystole
* No chronic active hepatitis or cirrhosis requiring treatment except hepatitis virus carriers who do not need treatment
* No comorbidity of interstitial pneumonia and pulmonary fibrosis requiring treatment
* No other cancer requiring treatment except a malignant tumor curatively resected with no recurrence
* No severe psychiatric disorders including schizophrenia or dementia
* Cardiothoracic ratio < 60% by chest x-ray
* No history of severe drug allergy or allergy to polyoxyethylene castor oil (in some anesthetic drugs or muscle relaxants) or polysorbate 80
* Patients in whom nitroglycerin preparations are contraindicated are not eligible, including any of the following:

  * Severe hypotension (e.g., systolic blood pressure ≤ 80 mm Hg)
  * Angle-closure glaucoma
  * History of hypersensitivity to nitrate/nitrite ester drugs
* Not pregnant or nursing

PRIOR CONCURRENT THERAPY:

* No prior chemotherapy or radiotherapy

  * Pleurodesis is not considered chemotherapy
* At least 1 week since prior and no other concurrent nitric oxide donors (e.g., nitroglycerin)
* At least 1 week since prior and no concurrent calcium antagonists
* At least 1 week since prior and no concurrent drugs for erectile dysfunction that inhibit phosphodiesterase 5 (e.g., sildenafil citrate or vardenafil hydrochloride hydrate)
* More than 24 hours since prior and no concurrent administration of the following:

  * Antifungal azoles, including ketoconazole, miconazole, or itraconazole
  * Macrolides, including erythromycin or clarithromycin
  * Cyclosporines
  * Benzodiazepines, including diazepam, triazolam, or midazolam
  * Vitamin A
  * Steroid hormones, including ethinylestradiol
* No concurrent participation in another clinical trial

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2008-01; Primary Completion 2011-12 (Estimated)

PRIMARY OUTCOMES:
Tumor response rate

SECONDARY OUTCOMES:
Progression-free survival
Adverse event and its severity
Overall survival
Change in the plasma concentration of VEGF between before and after the three-day administration of nitroglycerin prior to the start of the administration of anticancer drugs in the first course of the treatment
Change in the number of endothelial progenitor cells in blood between before and after the three-day administration of nitroglycerin prior to the start of the administration of anticancer drugs in the first course of the treatment
Blood concentration of paclitaxel and carboplatin immediately and two hours after the administration of the anticancer drug (paclitaxel) in the first course of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Hiroyasu Yasuda, MD, PhD, Study Chair — Tohoku University; Akiko Takeuchi — Translational Research Center for Medical Innovation, Kobe, Hyogo, Japan
Locations (1):
- Kyoto University Hospital, Kyoto, Kyoto, Japan